CLINICAL TRIAL: NCT05922774
Title: Evaluation of Cervical Vestibular Evoked Myogenic Potentials in Recurrent and Persistant Benign Paroxysmal Positional Vertigo
Brief Title: Cervical Vestibular Evoked Myogenic Potentials in Recurrent and Persistant Benign Paroxysmal Positional Vertigo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ISIL TAYLAN CEBI, principal investigator, Haseki Training and Research Hospital
Other Study IDs: cVEMP in intractable BPPV
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Benign Paroxysmal Positional Vertigo; Cervical Vestibular Evoked Myogenic Potentials; Vestibular Function Tests; Saccule and Utricle
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with recurrent BPPV
  Interventions: Device: Cervical VEMP testing
- Group 2: Patients with non recurrent BPPV
  Interventions: Device: Cervical VEMP testing
- Group 3: Healthy controls
  Interventions: Device: Cervical VEMP testing

INTERVENTIONS:
Device: Cervical VEMP testing — cervical vestibular evoked myogenic potentials

SUMMARY:
The goal of this observational study is to compare the cervical vestibular evoked myogenic potentials in recurrent/persistant BPPV and nonrecurrent BPPV. Recurrent/persistant BPPV is considered as the patients who require more than one repositioning manuever for the resolution of symptoms and the recurrent cases in the first three months after the diagnosis.

The main question[s] it aims to answer are:

* Is there any difference between the cVEMP findings of diseased ears of recurrent and nonrecurrent BPPV cases?
* Is there any difference between the cVEMP findings of diseased ears and healthy ears of BPPV patients
* Is there any difference between the cVEMP findings of healthy ears of recurrent and nonrecurrent BPPV cases and healthy controls?

Patients with VNG confirmed BPPV will be recruited and CVEMP test will be performed before the therapeutic manuevers.

Control visits will be scheduled on the 7th day after the therateutic menuevers are performed.

Patients will be followed-up for 4 weeks after the resolution of symptoms. Researchers will compare recurrent (Group 1), nonrecurrent (group 2) BPPV patients and healthy controls (Group 3) to see if there is any difference between the cVEMP findings of two groups.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to ENT clinic with unilateral posterior or lateral canal BPPV for the first time

Exclusion Criteria:

* patients with bilateral BPPV
* patients with recurrent or resistant BPPV
* patients with spontaneous nystagmus
* vestibular or neurologic disorders other than BPPV
* patients who use medication which may affect the vestibular system or muscle tone
* cervical muscle disorders and ocular pathologies which may affect the VEMP results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18-65 years of age with first BPPV attack confirmed with VNG.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The comparison of cVEMP findings in normal controls and BPPV patients with nonrecurrent and recurrent BPPV symptoms after 4 week follow-up. | 13 weeks
  Patients with VNG confirmed BPPV will be recruited and CVEMP test will be performed before the therapeutic manuevers.
  Control visits will be scheduled on the 7th day after the therapeutic menuevers are performed.
  Patients will be followed-up for 4 weeks after the resolution of symptoms. Researchers will compare recurrent (Group 1), nonrecurrent (group 2) BPPV patients and healthy controls (Group 3) to see if there is any difference between the cVEMP findings of these groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karatas A, Yuce T, Cebi IT, Acar Yuceant G, Haci C, Salviz M. Evaluation of Cervical Vestibular-Evoked Myogenic Potential Findings in Benign Paroxysmal Positional Vertigo. J Int Adv Otol. 2016 Dec;12(3):316-320. doi: 10.5152/iao.2016.2170. Epub 2016 Aug 1. PMID 28031157
- [Background] Yetiser S, Ince D, Gul M. An analysis of vestibular evoked myogenic potentials in patients with benign paroxysmal positional vertigo. Ann Otol Rhinol Laryngol. 2014 Oct;123(10):686-95. doi: 10.1177/0003489414532778. Epub 2014 May 1. PMID 24789801
- [Background] Xu H, Liang FY, Chen L, Song XC, Tong MC, Thong JF, Zhang QQ, Sun Y. Evaluation of the utricular and saccular function using oVEMPs and cVEMPs in BPPV patients. J Otolaryngol Head Neck Surg. 2016 Feb 9;45:12. doi: 10.1186/s40463-016-0125-7. PMID 26857819
- [Background] Kim EJ, Oh SY, Kim JS, Yang TH, Yang SY. Persistent otolith dysfunction even after successful repositioning in benign paroxysmal positional vertigo. J Neurol Sci. 2015 Nov 15;358(1-2):287-93. doi: 10.1016/j.jns.2015.09.012. Epub 2015 Sep 5. PMID 26371697
- [Background] Vaduva C, Esteban-Sanchez J, Sanz-Fernandez R, Martin-Sanz E. Prevalence and management of post-BPPV residual symptoms. Eur Arch Otorhinolaryngol. 2018 Jun;275(6):1429-1437. doi: 10.1007/s00405-018-4980-x. Epub 2018 Apr 23. PMID 29687182